CLINICAL TRIAL: NCT05763797
Title: Developing a Culturally Relevant Supportive Care Program for Black Patients Dealing With Advanced Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-1015; NCI-2023-01995 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 1 (individual interview) (Experimental): Participants will be interviewed
  Interventions: Behavioral: Individual Interview; Behavioral: Meditation Exercise
- Aim 2 (supportive care program) (Experimental): Participants will be assigned to one of two groups
  Interventions: Behavioral: Individual Interview; Behavioral: Meditation Exercise
- Aim 3 (supportive care program) (Experimental): Participants will be assessed regarding their program participation
  Interventions: Behavioral: Individual Interview; Behavioral: Meditation Exercise

INTERVENTIONS:
Behavioral: Individual Interview — Group 1, participant will be in a supportive care program with other Black cancer patients in which you will practice meditation.
  Group 2, participate will be in a supportive care program with other Black cancer patients that focuses on coping with cancer.
  Participants will be asked to participate weekly sessions for 4 weeks (that is a total of 4 sessions) and each session will last about 60 minutes. Both groups will be delivered via Zoom (a web-based videoconferencing service) and led by a master's-level interventionist.
Behavioral: Meditation Exercise — Group 1, participant will be in a supportive care program with other Black cancer patients in which you will practice meditation.
  Group 2, participate will be in a supportive care program with other Black cancer patients that focuses on coping with cancer.
  Participants will be asked to participate weekly sessions for 4 weeks (that is a total of 4 sessions) and each session will last about 60 minutes. Both groups will be delivered via Zoom (a web-based videoconferencing service) and led by a master's-level interventionist.

SUMMARY:
To determine the feasibility of implementing a culturally adapted mind-body intervention (Meditation-Based Support-Adapted; MBS-A) as a supportive care strategy in Black patients diagnosed with a stage III-IV solid malignancy. To target the specific needs of Black advanced cancer patients, we will first conduct formative research that includes quantitative surveys and in-depth interviews of patients and their primary caregivers. The purpose of this formative research is to determine the intervention format for the MBS-A program (family- vs group-based) that promises the greatest likelihood of success and to solicit input on the original MBS intervention regarding content that needs adaptation. Once the intervention format is determined and content adapted, we will conduct a pilot randomized controlled trial (RCT) to examine the feasibility of the MBS-A intervention vs. a dose-matched attention control (AC) group receiving a psychoeducation intervention.

DETAILED DESCRIPTION:
Primary Objectives:

The purpose of this RCT is to thoroughly determine the feasibility of the overall RCT design as well as specific intervention procedures in this underserved population to inform if a large efficacy trial is warranted. Our results will lead to future NIH R01 applications in which efficacy and mechanisms of the interventions will be tested using fully powered samples of Black patients with advanced cancer including multicenter trials. The long-term goal is to establish the effectiveness of the MBS-A intervention and widely disseminate the intervention. Ultimately, the intervention is intended to improve cancer control and reduce the double disparity in this underserved patient population.

We propose the following specific aims:

1. Systematically and culturally adapt a meditation-based support intervention (MBS-A) and finalize the intervention components and delivery format that meet the needs of Black patients with advanced cancer.
2. Identify the feasibility of conducting a supportive-care RCT in Black patients with advanced cancer as determined by recruitment and retention rates, randomization and blinding procedures, and intervention delivery.
3. Identify the feasibility of implementing the MBS-A and AC interventions as determined by session attendance, intervention acceptability, and treatment fidelity.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1, in order to be eligible to participate in this study, a patient must meet all of the following criteria:

* Self-identifies as Black/African American
* Is ≥18 years old
* Was diagnosed with a stage III-IV solid tumor
* Is able to provide informed consent

For Aims 2 and 3, in order to be eligible to participate in this study, a patient must meet all of the following criteria:

* Self-identifies as Black/African American
* Is ≥18 years old
* Was diagnosed with a stage III-IV solid tumor
* Is on active treatment (any line)
* Has an ECOG performance status of ≤2
* Has access to the internet
* Is able to provide informed consent

For Aims 2 and 3, if a family-based intervention is selected as the program format, a patient must meet the additional following criterion:

• Has a family caregiver (e.g., spouse, adult child) with whom they currently reside

Also, if a family-based intervention is selected as the program format, a caregiver must meet all of the following criteria:

* Is ≥18 years old
* Has access to the internet
* Is able to provide informed consent

Exclusion Criteria:

For Aim 1, there are no exclusion criteria.

For Aims 2 and 3, a patient who meets any of the following criteria will be excluded from participation in this study:

* Is pregnant
* Has cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team
* Participated in in the Aim 1 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory-Score Scale | through study completion; an average of 1 year.
  MD Anderson Symptom Inventory, which consists of 13 core items assessing symptom severity and 6 items assessing symptom interference with daily living.71,72 If the family-based format is selected, patients and caregivers will complete the form as it applies to their own symptoms as well as their perceptions of each other's symptoms.73
  MD Anderson Symptom Inventory-Score Scale "at its worst" using 0-10 numerical rating scales with 0 = "not present" and 10 = "as bad as you can imagine."

CONTACTS AND LOCATIONS:
Overall Officials: Dalnim Cho, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org